CLINICAL TRIAL: NCT01891097
Title: Combined Electroacupuncture and Auricular Acupuncture for Persistent Insomnia: A Randomized Controlled Trial of Dose-Response Effect
Brief Title: Combined Electroacupuncture and Auricular Acupuncture for Persistent Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Dr. Chung Ka-Fai, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACUP-005
Record Dates: First submitted 2013-06-20; First posted 2013-07-02 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Insomnia
Keywords: Insomnia; Acupuncture; Electroacupuncture; Aricular acupuncture; Randomized Clinical Trial; Traditional Chinese Medicine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Acupuncture Therapy; Acupuncture, Ear; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acupuncture (Active Comparator): Patients will be treated at bilateral Ear Shenmen, Sishencong EX-HN1, Anmian, Neiguan PC6, Shenmen HT7, Sanyinjiao SP6, and unilateral Yintang EX-HN3 and Baihui GV20. Acupuncture treatment will be performed by a registered Chinese medicine practitioner. "De qi"(an irradiating feeling considered to be indicative of effective needling) is achieved if possible. An electric-stimulator (ITO ES160, Japan) is connected to these needles to give an electric-stimulation in continuous wave, frequency of 4 Hz, 0.4 ms square wave pulses and constant current. Surgical tape or hair pin will be adhered to the needles.The needles will be left for 30 min and then removed. Acupuncture treatment will consist of three sessions per week for 3 consecutive weeks.
  Interventions: Procedure: Acupuncture
- Acupuncture plus auricular acupuncture (Experimental): Subjects will be treated with electroacupuncture plus auricular acupuncture for 3 weeks. The acupuncture regimen, is the same as in electroacupuncture group. In additional to electroacupuncture, subjects will receive auricular acupuncture using borneol. The following 6 ear acupoints points will be selected: Ear Shenmen, Heart, Kidney, Liver, Spleen, Occiput, and Subcortex. In each treatment borneol crystals will be attached to the left or right side of the ear in alternation with adhesive plaster in each acupuncture treatment visit. Subjects will be asked to press the borneol crystals lightly for five minutes in the morning, afternoon and evening everyday and reminded them to remove the plaster and borneol crystals after 48 hours. We will check for skin irritation at each treatment visit.
  Interventions: Procedure: Acupuncture plus auricular acupuncture
- Waiting-list control (No Intervention): This group will receive no treatment. Subjects will be assessed at baseline and the 4th and 7th week; afterwards, they will be randomized to one of the other two groups in the ratio of 1:1.

INTERVENTIONS:
Procedure: Acupuncture plus auricular acupuncture — Acupuncture at bilateral Ear Shenmen, Sishencong EX-HN1 , Anmian , Neiguan PC6 , Shenmen HT7 , Sanyinjiao SP6 , and unilateral Yintang EX-HN3 and Baihui GV20. The needles will be left for 30 min and then removed. Acupuncture treatment will consist of three sessions per week for 3 consecutive weeks.
  Aricular acupuncture at Ear Shenmen, Heart, Kidney, Liver, Spleen, Occiput, and Subcortex.In each treatment borneol crystals will be attached to the left or right side of the ear in alternation with adhesive plaster in each acupuncture treatment visit. Subjects will be asked to press the borneol crystals lightly for five minutes in the morning, afternoon and evening everyday and reminded them to remove the plaster and borneol crystals after 48 hours.
  Other Names: Acupuncture; Electroacupuncture
  Arms: Acupuncture plus auricular acupuncture
Procedure: Acupuncture — Acupuncture at bilateral Ear Shenmen, Sishencong EX-HN1 , Anmian , Neiguan PC6 , Shenmen HT7 , Sanyinjiao SP6 , and unilateral Yintang EX-HN3 and Baihui GV20. The needles will be left for 30 min and then removed. Acupuncture treatment will consist of three sessions per week for 3 consecutive weeks.
  Other Names: Electroacupuncture
  Arms: Acupuncture

SUMMARY:
This is a randomized controlled trial to evaluate the clinical efficacy of combined electro-acupuncture and auricular acupuncture for persistent Iinsomnia in the adult population in Hong Kong.

DETAILED DESCRIPTION:
Combined electro-acupuncture and auricular acupuncture is potential to be an alternative treatment for primary insomnia. The purpose of this study is to evaluate the clinical effectiveness of combined electroacupuncture and auricular acupuncture on persistent insomnia. This is a randomized double-blinded controlled trial. Patients will be randomly assigned to the electro-acupuncture group, the electro-acupuncture plus auricular acupuncture group or the waitlist controlled group. Patients will be put into groups and then compared.The chance of getting into each group is 3:3:1.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Hong Kong residents
* Ethnic Chinese
* Meet the diagnosis criteria of presistent insomnia for at least 3 months according to Current Diagnostic and Statistical Manual of Mental Disorders (the proposed Fifth Edition)
* Insomnia more than 3 nights per week for at least 3 months
* Willing to give informed consent
* Able to comply with trial protocol

Exclusion Criteria:

* Have a Hamilton Depression Rating Scale scores above 18
* Have sleep apnea or periodic limbs movement disorder detected by overnight polysomnography
* Have suicidal risk as assessed by the Hamilton Depression Rating Scale suicidal risk item
* Have current major depressive disorder, generalized anxiety disorders or panic disorder, manic or hypomanic episode, substance use disorders except caffeine and nicotine, organic mental disorder, schizophrenia or any other psychotic disorder
* Receiving psychotropic drugs with dosage changes in the last 4 weeks prior to screening, baseline or during the study
* Have valvular heart defects or bleeding disorders or were taking anticoagulant drugs
* Are pregnant, breast-feeding, or woman of childbearing potential not using adequate contraception
* Have any unstable psychiatric conditions or serious physical illnesses which are judged by the investigator to render unsuitable or unsafe
* Have infection or abscess close to the site of selected acupoints and in the investigator's opinion inclusion is unsafe
* Taking Chinese herbal medicine or over-the-counter drugs which are intending for insomnia within the last 2 weeks prior to baseline or during the study
* Any acupuncture or auricular acupuncture treatment during the previous 6 months prior to baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes of sleep parameters by subjective measures using sleep log | Baseline, 1-week posttreatment, 4-week posttreatment, and 13-week posttreatment
  We will measure sleep parameters (including sleep onset latency, sleep efficiency, total sleep time, times of wakening during sleep) by subjective measures using sleep log. The measure is a composite outcome measure consisting of multiple measures

SECONDARY OUTCOMES:
Change of self-rated sleep quality score measured by Insomnia Severity Index (ISI) questionnaire | Baseline, 1-week posttreatment, 4-week posttreatment, and 13-week posttreatment
Change of self-rated sleep quality score measured by the Pittsburgh Sleep Quality Index (PSQI) questionnaire | Baseline, 1-week posttreatment, 4-week posttreatment, and 13-week posttreatment
Change of anxiety and depression states measured by Hospital Anxiety and Depression Scale (HADS) | Baseline, 1-week posttreatment, 4-week posttreatment, and 13-week posttreatment
Change of subjects' functioning regarding work/study, social life and family measured by Sheehan Disability Scale (SDS) | Baseline, 1-week posttreatment, 4-week posttreatment, and 13-week posttreatment
Change of subjects' self-rated fatigue score measured by Multidimensional Fatigue Inventory (MFI) | Baseline, 1-week posttreatment, 4-week posttreatment, and 13-week posttreatment
Change of subjects' likeliness of dozing measured by Epworth Sleepiness Scale (ESS) | Baseline, 1-week posttreatment, 4-week posttreatment, and 13-week posttreatment
Change of subjects' sleep-related cognition measured by Dysfunctional Beliefs and Attitudes about Sleep (DBAS) | Baseline, 1-week posttreatment, 4-week posttreatment, and 13-week posttreatment
Change of subjects' sleep inhibitory behaviors measured by Sleep Hygiene Practice Scale (SHPS) | Baseline, 1-week posttreatment, 4-week posttreatment, and 13-week posttreatment
Change of subjects' credibility to the treatment measured by Credibility of treatment rating scale | Second and the last time of the treatment; 1-week posttreatment, 4-week posttreatment, and 13-week posttreatment
Change of sleep parameters (sleep onset latency, sleep efficiency, total sleep time, times of wakening during sleep) by objective measure - wrist actigraphy | Baseline, 1-week posttreatment, 4-week posttreatment, and 13-week posttreatment
  Sleep parameters include sleep onset latency, sleep efficiency, total sleep time, times of wakening during sleep. The measure is a composite outcome measure consisting of multiple measures
Change of serious adverse events measured by Serious Adverse Event (SAE) | 1-week posttreatment, 4-week posttreatment, and 13-week posttreatment
Change of potential adverse events related to acupuncture measured by Adverse Events Report Related to Acupuncture | 1-week posttreatment, 4-week posttreatment, and 13-week posttreatment

CONTACTS AND LOCATIONS:
Overall Officials: Ka-Fai Chung, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chung KF, Yeung WF, Ho FYY, Ng TK. Dysfunctional cognition regarding sleep as a mediator of outcome following acupuncture for insomnia. Acupunct Med. 2018 Jun;36(3):193-194. doi: 10.1136/acupmed-2017-011520. Epub 2018 Mar 22. No abstract available. PMID 29567667
- [Derived] Chung KF, Yeung WF, Yu BY, Leung FC, Zhang SP, Zhang ZJ, Ng RM, Yiu GC. Acupuncture with or without combined auricular acupuncture for insomnia: a randomised, waitlist-controlled trial. Acupunct Med. 2018 Feb;36(1):2-13. doi: 10.1136/acupmed-2017-011371. Epub 2017 Dec 11. PMID 29229613